CLINICAL TRIAL: NCT05429294
Title: Pyrotinib Combined With Trastuzumab and Albumin Paclitaxel in First-line Treatment of HER2-positive Advanced or Metastatic Breast Cancer, a Prospective, Single-arm, Multicenter, Phase II Study
Brief Title: Novel Double Target Therapy Combined With Chemotherapy in First-line Treatment of HER2+ Breast Cancer, MA-BC-II-038
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X-XJTU1AFLSY-93
Record Dates: First submitted 2022-06-18; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Pyrotinib combined with trastuzumab and albumin paclitaxel
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Patients with HER2-positive advanced/metastatic breast cancer are treated with pyrotinib combined with trastuzumab and albumin paclitaxel in the first-line setting.
  Other Names: Trastuzumab; Albumin paclitaxel

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of pyrotinib combined with trastuzumab and albumin paclitaxel in first-line treatment of HER2-positive advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years and ≤75 years.
* Pathologically confirmed diagnosis of Her2-positive advanced or metastatic breast cancer.
* ECOG 0 ~ 1.
* At least one measurable lesion according to RECIST 1.1.
* No prior anti-HER2 therapy and chemotherapy for MBC, and other anti-tumor therapy that the investigator considers to be excluded, and are permitted to undergo local therapy for local symptoms, such as radiotherapy for relief of bone pain.
* Patients with a disease-free interval of ≥12 months between the end of systemic therapy (except endocrine therapy) and tumor recurrence/metastasis after prior adjuvant/neoadjuvant systemic therapy are permitted.
* Life expectancy is not less than 12 weeks.
* hormone receptor status is known.
* Normal function of important organs, including heart, liver, lung, kidney and bone marrow.
* Volunteered to participate in the study, signed informed consent, had good compliance and was willing to cooperate with follow-up.

Exclusion Criteria:

* Patients with central nervous system metastasis.
* Inability to swallow, chronic diarrhea and intestinal obstruction, there are many factors that affect drug taking and absorption.
* Patients who had received radiotherapy, chemotherapy, surgical treatment (excluding local puncture) or molecular targeted therapy within 4 weeks prior to enrollment.
* Those who had received endocrine therapy within 2 weeks before enrollment.
* Tyrosine kinase inhibitors targeting HER2 (lapatinib, neratinib, pyrolitinib, etc.) have been used or are currently being used.
* Have used or are using T-DM1 before.
* Other malignancies within the past 5 years, excluding cured carcinoma in situ of the cervix, basal cell carcinoma of the skin or squamous cell carcinoma of the skin.
* The researchers judged those who were not eligible for systemic chemotherapy.
* Patients had undergone major surgical procedures or significant trauma in the 4 weeks prior to enrollment, or were expected to undergo major surgical treatment.
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B, hepatitis C (positive for hepatitis C antibodies and hcV-RNA higher than the detection limit for analytical methods) or co-infection with hepatitis B and C.
* History of any heart disease including :(1) angina pectoris; (2) arrhythmias requiring drug treatment or of clinical significance; (3) myocardial infarction; (4) heart failure; (5) Any other heart disease deemed unsuitable for the study by the investigator.
* Pregnant, lactating women, fertile women who tested positive for baseline pregnancy, or women of childbearing age who were unwilling to use effective contraception during the entire trial period.
* According to the judgment of the investigator, there are serious concomitant diseases (including but not limited to severe hypertension that cannot be controlled by drugs, severe diabetes, active infection, etc.) that seriously endanger patients' safety or affect patients' ability to complete the study.
* Known allergy to pyrotinib, trastuzumab, albumin paclitaxel or any excipient.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Concomitant use of CYP3A4 inhibitors or inducers or ongoing use of drugs that prolong QT interval.
* Known history of psychotropic substance abuse or drug abuse.
* Other serious physical or mental disorders or abnormalities in laboratory tests that may increase the risk of study participation or interfere with study results, and any other conditions that the investigator considers inappropriate for study participation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
PFS | during the procedure
  The length of the time during and after the treatment until disease progressed

SECONDARY OUTCOMES:
ORR | during the procedure
  The percent of patients who have CR or PR among all the patients enrolled
OS | during the procedure
  The the length of time from the enrollment to death

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Jin Yang, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No